CLINICAL TRIAL: NCT00957372
Title: Efficacy and Safety of BIA 2-093 as Adjunctive Therapy for Refractory Partial Seizures in a Double-blind, Randomized, Placebo-controlled, Parallel-group, Multicenter Clinical Trial
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate as Adjunctive Therapy for Refractory Partial Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-303
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Partial Epilepsy
Keywords: epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ESL 800 mg daily (Part I) (Experimental): ESL 800mg daily
  Interventions: Drug: eslicarbazepine acetate
- ESL 1200 mg daily (Part I) (Experimental): ESL 1200mg daily
  Interventions: Drug: eslicarbazepine acetate
- placebo (Part I) (Placebo Comparator): placebo
  Interventions: Drug: placebo (Part I)
- ESL - Open-label Extension (Part II) (Experimental): All patients were treated with only ESL during Part II.
  Interventions: Drug: ESL - Open-label Extension (Part II)

INTERVENTIONS:
Drug: eslicarbazepine acetate — oral tablet, 800 mg or 1200 mg once daily
  Other Names: Zebinix
  Arms: ESL 1200 mg daily (Part I); ESL 800 mg daily (Part I)
Drug: placebo (Part I) — once daily placebo comparator
  Arms: placebo (Part I)
Drug: ESL - Open-label Extension (Part II) — Part II was a 1-year open-label extension for patients who had completed Part I. Starting at 800 mg/day, the dosage could be titrated at 400 mg intervals down to a minimum of 400 mg/day or up to a maximum of 1200 mg/day
  Arms: ESL - Open-label Extension (Part II)

SUMMARY:
The primary objective was to evaluate the efficacy of eslicarbazepine acetate (ESL) administered once daily at 1200 mg or 800 mg, compared with placebo as adjunctive therapy in patients with refractory partial epilepsy over a 12-week maintenance period.

DETAILED DESCRIPTION:
This was a phase III, 2-part multicenter study. Part I was an 26-week parallel-group, randomized, placebo-controlled design consisting of an 8 week baseline period, a 2 week double-blinded titration period, 12 week maintenance period, and a 4 week tapering-off period. After completing the baseline period, patients were randomized in a 1:1:1 ratio to 1 of the 2 ESL daily dose levels (1200 or 800 mg) or placebo.

Part II was a 1-year open-label extension for patients who had completed Part I. Starting at 800 mg/day, the dosage could be titrated at 400 mg intervals down to a minimum of 400 mg/day or up to a maximum of 1200 mg/day. Patients who completed Part II could participate in a study extension and continue treatment with ESL until marketing authorization is obtained or clinical development is discontinued, with visits scheduled at the discretion of the investigator but at least every 6 months.

Results from Part I & II were presented in two separate reports.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent signed by patient
* aged 18 years or more
* documented diagnosis of simple or complex partial seizures with or without secondary generalisation since at least 12 months prior to screening
* at least 4 partial seizures in each 4 week period during the last 8 weeks prior to screening, currently treated with 1 or 2 AEDs (any except oxcarbazepine and felbamate), in a stable dose regimen during at least 2 months prior to screening (patients using vigabatrin should have been on this medication for at least 1 year with no deficit in visual field identified)
* excepting epilepsy, patient is judged to be in general good health based on medical history, physical examination and laboratory tests
* post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation; in case of woman of childbearing potential, patient must present a serum beta-hCG test consistent with a non-gravid state and agree to remain abstinent or use reliable contraception (oral contraception should be combined with a barrier method)

Exclusion Criteria:

* only simple partial seizures with no motor symptomatology (classified as A2-4 according to the International Classification of Epileptic Seizures) that are not video-EEG documented
* primarily generalised epilepsy
* known rapid progressive neurological disorder; history of status epilepticus or cluster seizures (i.e., 3 or more seizures within 30 minutes) within the 3 months prior to screening
* seizures of psychogenic origin within the last 2 years
* history of schizophrenia or suicide attempt
* currently on or with exposure to felbamate or oxcarbazepine more within one month of screening
* using benzodiazepines on more than on an occasional basis (except when used chronically as AED)
* previous use of ESL or participation in a clinical study with ESL
* known hypersensitivity to carbamazepine, oxcarbazepine or chemically related substances
* history of abuse of alcohol, drugs or medications within the last 2 years
* uncontrolled cardiac, renal, hepatic, endocrine, gastrointestinal, metabolic, haematological or oncology disorder
* second or third-degree atrioventricular blockade not corrected with a pacemaker
* relevant clinical laboratory abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2004-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil-Nagel, MD, Principal Investigator — Hospital Ruber Internacional La Masó 38, Mirasierra 28034 Madrid, Spain; Jose Lopes-Lima, MD, Principal Investigator — Hospital Santo António Largo Prof. Abel Salazar, 4099-001 Porto, Portugal
Locations (1):
- Bial - Portela & Cª, S.A., S. Mamede Do Coronado, Portugal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened at 39 sites in 3 countries.
  STUDY DATES:
  PART I: from: 14 Dec 2004 to: 19 Jan 2007 PART II: from 21 June 2005 to 22 January 2008
Pre-assignment Details: The duration of Part I was 26 weeks, including the 8-week baseline period. After completing the baseline period, patients were randomized in a 1:1:1 ratio to 1 of the 2 ESL daily dose levels (1200 or 800 mg) or placebo.Part II was a 1-year open-label extension for patients who had completed Part I
Groups:
- ESL 1200mg Daily: ESL 1200mg daily
  eslicarbazepine acetate : oral tablet, 800 mg or 1200 mg once daily
- ESL 800mg Daily: ESL 800mg daily
  eslicarbazepine acetate : oral tablet, 800 mg or 1200 mg once daily
- Placebo: placebo
  placebo : once daily placebo comparator
- Open-label Extension (Part II): Starting at 800 mg/day, the dosage could be titrated at 400 mg intervals down to a minimum of 400 mg/day or up to a maximum of 1200 mg/day.
Period: PART I
Arm/Group | ESL 1200mg Daily | ESL 800mg Daily | Placebo | Open-label Extension (Part II)
Started | 80 | 85 | 88 | 0
Safety Population | 80 | 85 | 87 | 0
Intention-to-Treat Population | 77 | 84 | 84 | 0
Per-Protocol Population | 35 | 47 | 51 | 0
Randomized But Not Treated | 0 | 0 | 1 | 0
Completed | 80 | 85 | 87 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Period: PART II
Arm/Group | ESL 1200mg Daily | ESL 800mg Daily | Placebo | Open-label Extension (Part II)
Started | 0 | 0 | 0 | 194
Safety Population | 0 | 0 | 0 | 194
Intention-to-treat (ITT) Population | 0 | 0 | 0 | 191
Per-Protocol Population | 0 | 0 | 0 | 108
Completed | 0 | 0 | 0 | 150
Not Completed | 0 | 0 | 0 | 44
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 8
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Not Know | 0 | 0 | 0 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 10
Not completed — Patient non-compliance | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESL 1200mg Daily | ESL 800mg Daily | Placebo | Total
Number analyzed (Participants) | 80 | 85 | 88 | 253
Age, Customized [Number; unit: participants]
  <=18 years | 2 | 2 | 2 | 6
  Between 18 and 65 years | 76 | 82 | 83 | 241
  >=65 years | 2 | 1 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 45 | 140
  Male | 35 | 35 | 43 | 113

OUTCOME MEASURES:

1. Primary Outcome: Seizure Frequency
Description: The primary efficacy endpoint is the natural log transformation of the seizure frequency per 4 weeks. The primary efficacy analysis was based on results for the ITT population during the 12-week maintenance period. Seizure frequency was compared between each active treatment group and the placebo group using an ANCOVA model with treatment as a factor and seizure frequency as a covariate
Time Frame: 12 weeks
Population: The primary efficacy analysis was based on the ITT population.The intent-to-treat (ITT) population included all randomized patients with at least one dose of investigational product and at least one post-baseline seizure frequency assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: ln (Seizures) per 4 weeks
Groups:
- Placebo: Placebo tablets matching the 400 and 600 mg active substance tablets were supplied.
- ESL 800 mg: 400 mg active substance tablets were supplied
- ESL 1200 mg: 400 and 600 mg active substance tablets were supplied
Arm/Group | Placebo | ESL 800 mg | ESL 1200 mg
Number analyzed (Participants) | 84 | 84 | 77
ln (Seizures) per 4 weeks | 7.3 [6.3 to 8.5] | 5.7 [4.9 to 6.7] | 5.5 [4.6 to 6.5]

2. Primary Outcome: PART II: Nº of Treatment-Emergent Adverse Events (TEAE)
Description: The primary objective for Part II of the study was to evaluate the safety and tolerability of eslicarbazepine acetate (ESL, BIA 2-093) at doses titrated to an efficacy or safety endpoint over a 1-year open-label period. Safety assessments were based primarily on AEs (Number of participants with at least one treatment-emergent adverse events are reported); assessment of AEs was based on treatment relatedness, action taken on study drug, outcome, and causality.
Time Frame: 1-year
Population: There was no sample size estimate for Part II. Part II was a 1-year open-label extension for patients who had completed Part I and was willing to continue treatment in Part II.
Measure: Number; unit: participants
Groups:
- TEAE; TEAE With Onset Within the First 4 Weeks of Part II; TEAE With Onset After the First 4 Weeks of Part II; Treatment-related Treatment-emergent Adverse Event; TEAE Leading to Discontinuation From the Study; Treatment Emergent Serious Adverse Event; TEAE Leading to Death: Starting at 800 mg/day, the dosage could be titrated at 400 mg intervals down to a minimum of 400 mg/day or up to a maximum of 1200 mg/day.
Arm/Group | TEAE | TEAE With Onset Within the First 4 Weeks of Part II | TEAE With Onset After the First 4 Weeks of Part II | Treatment-related Treatment-emergent Adverse Event | TEAE Leading to Discontinuation From the Study | Treatment Emergent Serious Adverse Event | TEAE Leading to Death
Number analyzed (Participants) | 194 | 194 | 194 | 194 | 194 | 194 | 194
participants | 112 | 40 | 94 | 66 | 9 | 11 | 2

ADVERSE EVENTS:
Time Frame: Overall study
Groups:
- Open-label Extension (Part II): ESL dose taken; Starting at 800 mg once daily, the dosage could be titrated at 400 mg intervals down to a minimum of 400 mg once daily or up to a maximum of 1200 mg once daily.
Arm/Group | Placebo | ESL 800 mg | ESL 1200 mg | Open-label Extension (Part II)
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/85 | 1/80 | 11/194
Other Adverse Events (participants affected / at risk) | 31/87 | 41/85 | 57/80 | 80/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=87) | ESL 800 mg (N=85) | ESL 1200 mg (N=80) | Open-label Extension (Part II) (N=194)
CEREBELLAR SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RHEUMATOID NODULES (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUSPECTED HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTION URINARY HYPONATREMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTROCYTOMA REFERS TO TUMORAL RELAPSE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THIRD GRADE BURN ON RIGHT ARM (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPILEPTIC STATUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POLYTRAUMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL HEMATOMA DUE TO HYSTERECTOMY COMPLICATIONS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CRANIAL TRAUMA - POLYCONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRANSITORY ISQUEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=87) | ESL 800 mg (N=85) | ESL 1200 mg (N=80) | Open-label Extension (Part II) (N=194)
Dizziness (Nervous system disorders) | 9 (9) | 16 (16) | 24 (24) | 33 (33)
Somnolence (Nervous system disorders) | 8 (8) | 11 (11) | 11 (11) | 19 (19)
Headache (Nervous system disorders) | 10 (10) | 5 (5) | 8 (8) | 17 (17)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 8 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 6 (6) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other